CLINICAL TRIAL: NCT06776471
Title: Clinical Evaluation of Two Different Pit and Fissure Sealants Used in Teeth Affected by Molar Incisor Hypomineralization
Brief Title: Clinical Evaluation of Two Different Pit and Fissure Sealants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-121
Record Dates: First submitted 2024-12-30; First posted 2025-01-15 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Pit and Fissure Sealants; Molar Incisor Hypomineralization
MeSH Terms: conditions — Van der Woude syndrome; Molar Hypomineralization

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Application of resin composite fissure sealant (Experimental): The occlusal surface will be etched with 37% phosphoric acid for 30 seconds, rinsed, and air dried until the enamel becomes opaque. Low-viscosity fluoride containing resin-based fissure sealant will be applied to the etched enamel surface. All applied fissure sealants will be polymerized using a light device. Finally, occlusion control will be performed on fissure sealants with articulation paper.
  Interventions: Other: Resin-based flowable filling material
- Application of self adhesive flowable composite fissure sealant (Active Comparator): The occlusal surface will be etched with 37% phosphoric acid for 30 seconds, the surface will be rinsed and air dried until an opaque appearance is achieved on the enamel.The occlusal surface self adhesive flowable composite will be applied in one step. All applied fissure sealants will be polymerized using a light device. Finally, occlusion control will be performed on fissure sealants with articulation paper.
  Interventions: Other: Resin-based flowable filling material

INTERVENTIONS:
Other: Resin-based flowable filling material — Preventive restoration

SUMMARY:
It is planned to include girls and boys between the ages of 6-12 who apply to Başkent University Faculty of Dentistry, Pediatric Dentistry Clinic for routine dental examination. Informed and written consent will be obtained from the parents of each participating child. In teeth planned to undergo treatment, molar ıncisor hypomineralization diagnosis will be made primarily in the presence of limited opacities/enamel fracture after eruption in at least one first permanent molar according to European Academy of Paediatric Dentistry criteria. In teeth diagnosed with molar ıncisor hypominerlization, tooth surfaces will be cleaned with a slow-speed rotary brush and dried with air before the evaluations to be made using the ICDAS II index. Early enamel caries lesions will be assessed by visual examination.

The decayed, missing, filled teeth of the patients will be assessed according to the World Health Organization assessment criteria. The groups will be double-blind randomized as conventional fissure sealant (n=63) and self-adhesive flowable composite (n=63): Group I (acid+resin-based fissure sealant) will be etched with 37% phosphoric acid for 30 seconds, the surface will be rinsed and air dried until an opaque appearance is achieved on the enamel. Low-viscosity fluoride containing resin based fissure sealant will be applied to the etched enamel surface. Group II (self-adhesive flowable composite); self adhesive flowable composite will be applied in one step. All applied fissure sealants will be polymerized using a light device. Finally, occlusion control will be performed on fissure sealants with articulation paper.The Schiff Cold Air Sensitivity Scale will be used to assess the presence of hypersensitivity in the affected teeth by applying the air-water spray perpendicular to the occlusal surface of the tooth from a distance of 1 cm for 1 second. Clinical evaluation of fissure sealants will be performed at 1, 3, 6 and 12 months using modified . Sealants that receive "Alpha" or "Bravo" scores for all criteria (anatomical form, marginal adaptation, surface texture, marginal color change, retention and secondary caries) will be classified as successful; while "Charlie" scores received from one or more of the United States Public Health Service criteria will be evaluated as failure.

DETAILED DESCRIPTION:
According to the results of this study, if successful results can be obtained from self adhesive flowable composites used as fissure sealants in molar incisor hypomineralized teeth during the 12 month follow up period, it will be possible to shorten the time spent at the patient's bedside by reducing the procedure steps during dental treatment and to increase patient comfort. In addition, depending on the results obtained, self-adhesive flowable composites with different contents will be evaluated with further studies and a pioneering step will be taken for their routine use as fissure sealants with longer clinical life.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 6-12 years with at least two fully erupted permanent first molars diagnosed with molar ıncisor hypomineralization according to the European Academy of Paediatric Dentistry criteria.
* Hypomineralized first molars with enamel defects according to early lesions

Exclusion Criteria:

* Ongoing orthodontic treatment
* Uncooperative child during dental treatment
* Teeth with advanced lesions, existing restorations, fluorosis, or enamel malformation due to syndromic causes
* Presence of pulpal symptoms

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-11-18 (Estimated); Study Completion 2025-12-18 (Estimated)

PRIMARY OUTCOMES:
Using United States Public Health Service criteria | up to 12 month
  There is no clinical study on the use of self-adhesive flowable composites as fissure sealants in teeth with molar incisor hypomineralization. Therefore, this study contributes to the literature. In this study, it is anticipated that the use of self-adhesive flowable composites will increase as they show similar clinical success to traditional fissure sealants at the end of their 12-month clinical life. Clinical evaluation of fissure sealants will be performed at 1, 3, 6 and 12 months using modified United States Public Health Service criteria. Sealants receiving "Alpha" or "Bravo" scores for all criteria (anatomical form, marginal adaptation, surface texture, marginal discoloration, retention and secondary caries) will be classified as successful, while a "Charlie" score for one or more of the United States Public Health Service criteria will be considered as failure.

SECONDARY OUTCOMES:
Using The Schiff Cold Air Sensitivity Scale test | 12 month
  The Schiff Cold Air Sensitivity Scale will be used to assess the presence of hypersensitivity in the affected teeth by applying the air-water spray perpendicular to the occlusal surface of the tooth from a distance of 1 cm for 1 second. When evaluating this test, the patient will receive a minimum score of 0 and a maximum score of 3. The patient's response will be recorded as follows: 0 = the person does not respond to the stimulus; 1 = the person does not respond to the stimulus but feels the stimulus is painful; 2 = the person responds to the air stimulus and moves away from the stimulus, and 3 = the person responds to the air stimulus, moves away from the stimulus, and requests that the stimulus stop immediately.

CONTACTS AND LOCATIONS:
Overall Officials: Simge POLAT, Lecturer, Principal Investigator — Baskent University
Locations (1):
- Başkent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No